CLINICAL TRIAL: NCT03443583
Title: Prospective Randomized Clinical Trial on the Survival and Quality of Survival of Lithium Disilicate Posterior Partial Crowns Bonded Using Immediate or Delayed Dentin Sealing a 3- Year Follow up
Brief Title: Immediate and Delayed Dentin Sealing Effect on Partial Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Carline van den Breemer, Principal Investigator, University Medical Center Groningen
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: NL45130
Record Dates: First submitted 2018-02-18; First posted 2018-02-23 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Adhesion; Tooth; Crown; Luting; Immediate Dentin Sealing
MeSH Terms: conditions — Tissue Adhesions

STUDY DESIGN:
Intervention Model Description: A split mouth clinical trial comparing ceramic restorations cemented with either IDS or DDS after one year of three years of clinical service.
Who Masked: Participant
Masking Description: Only the participant does not know which treatment is used on which teeth. The care provider and investigator have to know because different treatment protocol steps that have to be taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Immediate Dentin Sealing or Delayed Dentin Sealing — The main difference between the IDS and DDS technique lies in the fact that in IDS, a thin layer of bonding resin is applied immediately after tooth preparation and prior to impression taking, whereas in DDS this layer is applied immediately before cementation of the restoration.

SUMMARY:
Immediate Dentin Sealing as an adjunct to adhesive cementation of all ceramic restorations is proposed and executed in several studies, but there is very limited evidence to support its effectiveness. It is presumed that IDS both reduces postoperative sensitivity and increases the bond strength to dentin as compared to DDS.

DETAILED DESCRIPTION:
Micromechanical and chemical retention of ceramic fixed prosthesis to tooth structure introduced minimal invasive preparation to dentistry. As a result, biomechanically or aesthetically compromised teeth can be restored at a lower biological price, saving sound tooth tissues. A slow but steady (mind) shift from full metal and metal-ceramic restorations that require conventional cementation and substantial tooth loss (Edelhoff en Sorensen, 2002) to less destructive partial all ceramic restorations that require adhesive cementation is seen in the clinical field.

The clinical success of ceramic restorations relies heavily on the quality of their adhesion to dentin, which remains a clinical challenge to date. Improvements in this field over the years have brought about better cements and more effective methods to condition both substrates and teeth.

Immediate Dentin Sealing (IDS) is a technique that presumably improves adhesion of ceramic fixed prosthesis to tooth structure which results in a better marginal adaptation to dentin and less postoperative sensitivity compared to conventional adhesive cementation, also referred to as Delayed Dentin Sealing (DDS).(Pashley et al, 1992; Paul en Scharer, 1997; Magne et al, 2005; Magne et al, 2007; Breschi et al, 2008; Lee en Park, 2009). The main difference between the IDS and DDS technique lies in the fact that in IDS, a thin layer of bonding resin is applied immediately after tooth preparation and prior to impression taking, whereas in DDS this layer is applied immediately before cementation of the restoration. At first glance this may appear a minor difference, but it is presumed to be of major clinical importance. The effectiveness of IDS is studied as an adjunct to conventional adhesive cementation of ceramic indirect restorations. A split mouth clinical trial comparing ceramic restorations cemented with either IDS or DDS after one year of clinical service is executed. For each patient two all ceramic indirect restorations are made. One is cemented by means of DDS (control group) and the other one is cemented by means of IDS (experimental group). Clinical evaluation is performed shortly after cementation and after 1 and 3 year(s) of clinical function.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be over 18 years of age, in reasonable to good general health, as expressed by an ASA-score I or II (de Jong and Abraham-Inpijn, 1994).This ASA-score is already known before participation, due to regular check-ups;
* Patients should have an indication for at least two indirect ceramic restorations on vital teeth.

Exclusion Criteria:

* ASA-score III or higher;
* Hypersensitivity of the tooth which has to be restorated. This is measured before inclusion. (Is measured with a cotton pallet and cold spray which are hold to the tooth. If the tooth is painful and is doesn't relief from pain quickly the tooth is hypersensitive)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Survival | 3 year
  Survival of the restorations

SECONDARY OUTCOMES:
Quality of the restorations | 3 year
  Criteria according to Hickel and USPHS

IPD SHARING:
Plan to Share IPD: No